CLINICAL TRIAL: NCT01054703
Title: Clinical Evaluation of the Safety and Feasibility of the Ethmoid Sinus Spacer and Access System With Drug (SPACER)
Brief Title: Clinical Evaluation of the Ethmoid Sinus Spacer
Acronym: SPACER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim assessment performed after 14 patients provided evidence that further enrollment was not required to achieve intended endpoints of the study.
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR02082
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2010-02-24 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Sinusitis, Chronic Rhinosinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ethmoid Sinus Spacer placement (Experimental): Ethmoid Sinus Spacer and Access System used for the local delivery of Kenalog-40
  Interventions: Device: Ethmoid Sinus Spacer

INTERVENTIONS:
Device: Ethmoid Sinus Spacer — Ethmoid Sinus Spacer and Access System used for the local delivery of Kenalog-40
  Other Names: Acclarent Ethmoid Sinus Spacer and Access System

SUMMARY:
Evaluation of treatment of the ethmoid sinuses with the Ethmoid Sinus Spacer and Access system

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 years old
2. Both male and female
3. Ethmoid disease on CT scan
4. At least one non-ethmoid sinus requiring treatment
5. Failed medical management and symptomatic

Exclusion Criteria:

1. Previous ethmoid surgery
2. Not sufficient room for placement of Spacer
3. Patient requires septoplasty
4. Has received steroid treatment with in 2 weeks
5. Extensive sinonasal osteoneogenesis preventing device placement
6. Sinonasal tumors or obstructive lesions
7. History of facial trauma that distorts sinus anatomy
8. Asthmatic patients with aspirin sensitivity
9. Pregnant or lactating females

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2007-11-01 (Actual); Study Completion 2007-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Kuhn, MD, Principal Investigator — Georgia Nasal and Sinus Institute
Locations (1):
- Georgia Nasal and Sinus Institute, Savannah, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ethmoid Sinus Spacer Placement
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ethmoid Sinus Spacer Placement
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Adverse Events at the Time of the Procedure and Cumulatively up to 6 Weeks Post-implant
Time Frame: Procedural and 6 weeks post-implant
Measure: Number; unit: participants
Arm/Group | Ethmoid Sinus Spacer Placement
Number analyzed (Participants) | 14
participants | 1

2. Secondary Outcome: Efficacy: Improvement in Ethmoid Sinus Health as Demonstrated by CT Scan and Quality-of-life Measures
Time Frame: 1 wk, 2wk, 4wk, 6wk
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ethmoid Sinus Spacer Placement
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ethmoid Sinus Spacer Placement (N=14)
epistaxis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator shall not issue or disseminate any press release or statement, nor initiate or cause to be initiated any communication of information regarding the clinical trial (written or oral) to the communications media or third parties without the prior written consent of Sponsor.